CLINICAL TRIAL: NCT01967615
Title: P2Y12 Inhibitors Utilization in Bifurcation and Chronic Total Occlusion PCI With Biologically Active Stents (P2BiTO) Registry
Brief Title: P2Y12 Inhibitors Utilization in Bifurcation and Chronic Total Occlusion PCI
Acronym: P2BiTO
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Raffaele De Caterina, MD/PhD, G. d'Annunzio University
Other Study IDs: P2BiTO13; 2013-100813 (Registry Identifier: P2BiTO)
Record Dates: First submitted 2013-10-17; First posted 2013-10-23 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Coronary Arteriosclerosis
Keywords: PCI,; CTO,; bifurcation,; clopidogrel,; prasugrel,; ticagrelor
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prasugrel and ticagrelor were both associated with a significant reduction in the risk of MACE in patients undergoing PCI for an ACS, mostly through a reduced stent thrombosis. The 1-year relative risk reduction (RRR) of definite of probable stent thrombosis in patients receiving a DES were fairly different in TRITON-TIMI 38 and PLATO trials. The incidence of "biologically active" stent (DES or BVS) thrombosis is largely variable according to different lesion settings. We aim to verify the translation of the postulated different reduction in thrombosis rate among various P2Y12 inhibitors (clopidogrel, prasugrel and ticagrelor) in a high-risk setting such as the PCI with DES or BVS in CTO and bifurcating lesions.

DETAILED DESCRIPTION:
All patients aged 18-80 who underwent PCI of a CTO or bifurcating lesion (all Medina types, side branch ≥2 mm) with "biologically active stents" (DES or BVS) between January 2012 and december 2014 at participating centers will be deemed eligible to enter the registry.

In-hospital outcomes will be recorded; all patients discharged alive will be followed up with a telephone interview (minimum follow-up 6 months).

The primary end-point will be the occurrence of a cluster of major adverse cardiovascular events at 1 year:

1. Death from any cause.
2. Myocardial infarction.
3. Stent thrombosis, defined as definite, probable or possible following the Academic Research Consortium.

Sample size 3150 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years old
* PCI of a CTO or bifurcating lesion (all Medina types, side branch ≥2 mm) with "biologically active stents"

Exclusion Criteria:

-none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18-80 undergoing PCI of a CTO or bifurcating lesion (all Medina types, side branch ≥2 mm) with "biologically active stents" (DES or BVS) between January 2012 and december 2014 at participating centers will be deemed eligible to enter the registry.
Sampling Method: Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Death, Myocardial infarction, Stent Thrombosis | 30 months
  1. Death from any cause.
  2. Myocardial infarction, defined as an elevation of the creatine kinase MB fraction or cardiac troponins by a factor of 3 or more, or the development of new Q waves in 2 or more contiguous leads at surface ECG7. Levels of total creatine kinase and the creatine kinase MB fraction will be measured in all patients between 12 and 24 hours after PCI.
  3. Stent thrombosis, defined as definite, probable or possible3 following the Academic Research Consortium

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zimarino, MD, Principal Investigator — G. d'Annunzio University

REFERENCES:
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] Cannon CP, Harrington RA, James S, Ardissino D, Becker RC, Emanuelsson H, Husted S, Katus H, Keltai M, Khurmi NS, Kontny F, Lewis BS, Steg PG, Storey RF, Wojdyla D, Wallentin L; PLATelet inhibition and patient Outcomes Investigators. Comparison of ticagrelor with clopidogrel in patients with a planned invasive strategy for acute coronary syndromes (PLATO): a randomised double-blind study. Lancet. 2010 Jan 23;375(9711):283-93. doi: 10.1016/S0140-6736(09)62191-7. Epub 2010 Jan 13. PMID 20079528
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Steg PG, Harrington RA, Emanuelsson H, Katus HA, Mahaffey KW, Meier B, Storey RF, Wojdyla DM, Lewis BS, Maurer G, Wallentin L, James SK; PLATO Study Group. Stent thrombosis with ticagrelor versus clopidogrel in patients with acute coronary syndromes: an analysis from the prospective, randomized PLATO trial. Circulation. 2013 Sep 3;128(10):1055-65. doi: 10.1161/CIRCULATIONAHA.113.002589. Epub 2013 Jul 30. PMID 23900047
- [Background] Valenti R, Vergara R, Migliorini A, Parodi G, Carrabba N, Cerisano G, Dovellini EV, Antoniucci D. Predictors of reocclusion after successful drug-eluting stent-supported percutaneous coronary intervention of chronic total occlusion. J Am Coll Cardiol. 2013 Feb 5;61(5):545-50. doi: 10.1016/j.jacc.2012.10.036. Epub 2012 Dec 26. PMID 23273395
- [Background] Zimarino M, Corazzini A, Ricci F, Di Nicola M, De Caterina R. Late thrombosis after double versus single drug-eluting stent in the treatment of coronary bifurcations: a meta-analysis of randomized and observational Studies. JACC Cardiovasc Interv. 2013 Jul;6(7):687-95. doi: 10.1016/j.jcin.2013.03.012. Epub 2013 Jun 14. PMID 23769650
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Derived] Zimarino M, Briguori C, Amat-Santos IJ, Radico F, Barbato E, Chieffo A, Cirillo P, Costa RA, Erglis A, Gamra H, Gil RJ, Kanic V, Kedev SA, Maddestra N, Nakamura S, Pellicano M, Petrov I, Strozzi M, Tesorio T, Vukcevic V, De Caterina R, Stankovic G; EuroBifurcation Club. Mid-term outcomes after percutaneous interventions in coronary bifurcations. Int J Cardiol. 2019 May 15;283:78-83. doi: 10.1016/j.ijcard.2018.11.139. Epub 2018 Dec 2. PMID 30528620

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT01967615/Prot_SAP_000.pdf